CLINICAL TRIAL: NCT00002396
Title: A Phase I/II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerance, Pharmacokinetics, and Antiviral Activity of 9-[2-(R)-[[Bis[[(Isopropoxycarbonyl)- Oxy]Methoxy]Phosphinoyl]Methoxy]Propyl]Adenine Fumarate (PMPA Prodrug) in HIV-Infected Patients
Brief Title: The Safety and Effectiveness of PMPA Prodrug in HIV-Infected Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 283A; GS-97-901
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Adenine; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
To evaluate the safety of single and multiple doses (28 daily doses) of 9-[2-(R)-[[bis[[(isopropoxycarbonyl)- oxy]methoxy]phosphinoyl]methoxy]propyl]adenine fumarate (PMPA) prodrug administered orally to HIV-infected patients. To determine the pharmacokinetics of single and multiple doses of PMPA prodrug when administered orally to HIV-infected patients. To evaluate the anti-HIV activity of PMPA prodrug, as demonstrated by increases in CD4 cell counts and decreases in HIV RNA, when administered orally as a single dose and daily for 4 weeks to HIV-infected patients with CD4 cell counts of 200 or more cells/mm3.

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled study, a total of 60 patients are randomized to receive PMPA prodrug at 1 of 5 doses or matching placebo tablets.

Part A (Days 1-7): Patients receive a single dose of PMPA prodrug or matching placebo tablets administered orally followed by a 1-week observation period. Patients who complete Part A without a dose-limiting toxicity begin Part B.

Part B (Days 8-35): Patients receive either PMPA prodrug or matching placebo tablets administered orally qd for 4 weeks at the same dosage level administered in Part A.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection, as indicated by seropositivity for HIV infection (ELISA and Western blot), positive HIV culture, or positive plasma HIV RNA.
* CD4 cell count of 200 or more cells/mm3 within 28 days prior to study entry.
* Plasma HIV RNA of 10,000 or more copies/ml within 28 days of study entry.
* Minimum life expectancy of 12 months.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active, serious infections (other than HIV infection) that require parenteral antibiotic therapy. Patients should be considered recovered if at least 2 weeks have elapsed following the cessation of parenteral antibiotic therapy before enrollment.
* Active clinically significant medical problems including cardiac disease (e.g., symptoms of ischemia, congestive heart failure, or arrhythmia).
* Positive test for Hepatitis B surface antigen (HBsAg).
* Malignancy other than basal cell carcinoma or cutaneous Kaposi's sarcoma.

Prior Medication:

Excluded:

* Adefovir dipivoxil (bis-POM PMEA) for more than 14 days.

Within 2 weeks prior to entry:

* Antiretroviral therapy, including nucleoside analogues, nonnucleoside reverse transcriptase inhibitors, protease inhibitors, or investigational antiretroviral agents.
* Interferon (alpha, beta, or gamma) or interleukin (e.g., IL-2) therapy, aminoglycoside antibiotics, amphotericin B, cidofovir, diuretics, foscarnet, ganciclovir, itraconazole, fluconazole, ketoconazole (topical allowed), isoniazid, rifampin, rifabutin, clarithromycin, azithromycin, systemic chemotherapeutic agents, systemic corticosteroids, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and other investigational agents.

Risk Behavior:

Excluded:

Active drug or alcohol abuse as demonstrated by a positive screening test for drugs of abuse (except marijuana or drugs used for medical indications) or substance abuse considered sufficient to hinder patient compliance.

Patients who are receiving:

* Antiretroviral therapy, including nucleoside analogues, nonnucleoside reverse transcriptase inhibitors, protease inhibitors, or investigational antiretroviral agents. NOTE:
* Antiretroviral therapy may be started after completion of the Day 49 follow-up visit (i.e., not earlier than 14 days after completion of dosing).
* Interferon (alpha, beta, or gamma) or interleukin (e.g., IL-2) therapy, aminoglycoside antibiotics, amphotericin B, cidofovir, diuretics, foscarnet, ganciclovir, itraconazole, fluconazole, ketoconazole (topical allowed), isoniazid, rifampin, rifabutin, clarithromycin, azithromycin, systemic chemotherapeutic agents, systemic corticosteroids, other agents with significant nephrotoxic potential, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and other investigational agents.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - San Francisco Gen Hosp, San Francisco, California
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of Washington / AIDS Clinical Trial Unit, Seattle, Washington